CLINICAL TRIAL: NCT03263793
Title: High-intensity Group Vocal Exercise to Improve Laryngeal Function in Patients With Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-00323
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Parkinson Disease
Keywords: singing
MeSH Terms: conditions — Parkinson Disease | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral vocal training (Experimental): 12-week vocal training program will use maximum vocal function exercises targeting vocal deficits specific to Parkinson Disease.
  Interventions: Behavioral: Choral (group) singing therapy sessions

INTERVENTIONS:
Behavioral: Choral (group) singing therapy sessions — Choral (group) singing therapy sessions will be conducted once weekly and daily home practice exercises will be assigned. All vocal exercises are based on principles that have been successful in other intensive Parkinson Disease vocal exercise programs.

SUMMARY:
The overall goal of this T2 translational research project is to pilot an interdisciplinary high-intensity group singing program to improve speech and swallowing in patients with Parkinson's Disease (PD) and to explore the impact of this program on quality of life (QOL). This research has three specific aims: 1) Determine the effects of a high-intensity group vocal training program on vocal function and laryngeal structure; 2) Determine the transference of vocal training to laryngeal aspects of swallowing; 3) Determine the effect of patient-reported changes in Quality of Life (QOL) as the result of participation in a group vocal training program.

Twenty patients with Parkinson Disease will be recruited from the Fresco Institute for Parkinson's & Movement Disorders to participate in a 12-week vocal training program. The program will train participants using maximum vocal function exercises targeting vocal deficits specific to PD. Choral singing therapy sessions will be conducted once weekly with daily home practice exercises based on principles that have been successful in other intensive PD vocal exercise programs.

DETAILED DESCRIPTION:
Deterioration of speech and swallowing is a hallmark of Parkinson Disease (PD). There is emerging evidence that choral singing benefits people with PD across a range of modalities. Despite the increasing popularity of "Parkinson's choirs", rigorous study of these benefits is lacking. There is a large body of evidence that intense vocal training improves speech and communication for people with PD. However, the intense training places high demands on clinical and patient resources and, due to its individualized approach, lacks the potential psycho-social benefits of a group intervention.

It is hypothesized singing training program will increase vocal loudness, range of articulation, and prosodic variation during speech. Additionally, given existing evidence for neuroplastic transference of voice-related interventions to swallowing function, laryngeal components of swallowing function will also improve post-intervention. Finally, investigators expect to see improvements in patient-reported QOL measures corresponding with improved speech and laryngeal function and/or as the result of group interaction.

All participants will complete a standardized battery of assessment pre- and post- treatment including acoustic and aerodynamic assessment of voice, dynamic magnetic resonance imaging of speech and swallowing, and videofluoroscopic evaluation of swallowing. The outcome of this work will be a rigorous understanding of how choral singing therapy can positively impact the voice, swallowing function, and quality of life for patients with PD.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Stage One, Two or Three on the Hoehn and Yahr Staging of Parkinson's Disease
* Current swallowing severity of normal, mild, or moderate without aspiration
* Stable regimen of anti-PD medication for >30 days

Exclusion Criteria:

* Prior voice and/or swallowing therapy related to PD
* History of head and neck cancer
* History of oropharyngeal or laryngeal surgery
* Current or former smoker (quit < 5 years)

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-13 (Actual)

PRIMARY OUTCOMES:
Average speaking intensity (dB SPL) | 19 Weeks
  Tasks: Sustained phonation of /a/ at a comfortable pitch and loudness for 4 seconds; pitch glide throughout physiologic vocal range on /a/; standardized reading passage (CAPE-V sentences); 1-minute monologue in response to an emotionally neutral question; singing a standard song.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Johnson, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States